CLINICAL TRIAL: NCT05207761
Title: A Randomized, Open-label, 2-period, Parallel Group, Multiple-dose Phase 1 Study to Evaluate Drug-drug Interaction, Safety and Tolerability in Case of the Co-administration of D565 and D930, in Healthy Male Subjects
Brief Title: Study to Evaluate Drug-drug Interaction, Safety and Tolerability in Case of the Co-administration of D565 and D930
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A71_05DDI2114
Record Dates: First submitted 2022-01-04; First posted 2022-01-26 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): 1. Period 1: D565 7days
  2. Period 2: D565+D930 91days
  Interventions: Drug: D565; Drug: D930
- Sequence 2 (Experimental): 1. Period 1: D930 91days
  2. Period 2: D565+D930 7days
  Interventions: Drug: D565; Drug: D930

INTERVENTIONS:
Drug: D565 — Q.D. in both eye
Drug: D930 — T.I.D in both eye

SUMMARY:
This study is a randomized, open-label, 2-period, parallel group, multiple-dose phase 1 study to evaluate drug-drug Interaction, safety and tolerability in case of the co-administration of D565 and D930, in healthy male subjects

DETAILED DESCRIPTION:
To healthy male subjects of thirty-two (32), Investigational products are administered following treatments in each period

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults volunteers aged between 19 and 55 years old at the time of screening
2. Weight ≥ 55 kg, Calculated Body Mass Index(BMI) of 18.0 to 30.0 kg/m2

   * BMI = Weight(kg)/ Height(m)2
3. Individuals who sign an informed consent form and decide to participate in the study after being fully informed of the study prior to participation
4. Individuals who are suitable as a subject for this study at the discretion of the researcher as a result of screening tests such as examination, laboratory tests and questionnaires

Exclusion Criteria:

1. Individuals who have other clinically significant cardiovascular system, respiratory system, liver, renal, nervous system, endocrine system, blood-oncology, psychiatric disorders, urinary system or ophthalmic diseases or have a history
2. Individuals who satisfy the following items during the interview or examination

   * Individuals with a history of or sign or symptoms of a disease of the visual system
   * Individuals who had an ophthalmic surgery including for refractive correction surgery such as LASIK.
   * Individuals with corrected visual acuity of 20/40 or less
   * Individuals who have experienced side effects after wearing contact lenses or who have worn contact lenses within the last month
   * Individuals who have more than 21mmHg or less than 10mmHg on either side of the intraocular pressure test
   * Individuals who show abnormal findings in other ophthalmic examinations
3. Individuals who have a history of hypersensitivity to the active ingredient and component of the investigational drug, or to the drug in the same class as the active ingredient
4. Individuals with sitting systolic blood pressure ≥ 140 mmHg or ≤ 80 mmHg or sitting diastolic blood pressure ≥ 90 mmHg or ≤ 45 mmHg
5. Individuals with the following results at screening test

   * AST, ALT, γ-GT > 2x the upper limit of the normal range
   * Total bilirubin > 2.0 mg/dL
   * eGFR(CKD-EPI) < 60 mL/min/1.73m2
6. Individuals who continue to drink(over 21 units/week) within 1 month or cannot abstain from alcohol during the clinical trial period
7. Individuals who tested positive in an alcohol breath analysis
8. Individuals who continuously smoke within one month(including e-cigarettes, over 10 fees/day) or who cannot quit smoking during the clinical trial period;
9. Individuals who cannot restrict the intake of grapefruit or grapefruit-containing food from 3 days before administration of investigational drugs to the final pharmacokinetic blood sample collection
10. Individuals who tested positive for urine cotinine at screening test
11. Individuals who took ethical(ETC) or oriental medicine within 2 weeks or over the counter(OTC) within 1 week before the expected first dose
12. Individuals taking medication known to significantly induce or inhibit drug metabolizing enzymes within 1 month before the expected first dose
13. Individuals with a medical history of significant drug abuse or positive for abuse drug in urine test results at screening
14. Individuals who had been administered investigational product(s) of other clinical study within the 6 months prior to the first dose of this study
15. Individuals who donated whole blood within the 2 months, or donated blood components within 1 month, or received a blood transfusion with 1month prior to the first dose or plan to donate blood or transfusion during the clinical trial period
16. Individuals who are unable to use an appropriate medically approved method of contraception for themselves, their spouses, or partners during the entire clinical trial period and for at least 90 days after the last investigational drug administration and cannot donate sperm during this period
17. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss of D565(Sequence1) | 1day 0hour ~ 99day 0hour
  Area under the D565 concentration in blood-time curve from 0 to τ at steady state
AUCtau,ss of D930(Sequence1) | 8day 0hour ~ 99day 0hour
  Area under the D930 concentration in blood-time curve from 0 to τ at steady
AUCtau,ss of D565(Sequence2) | 96day 0hour ~ 99day 0hour
  Area under the D565 concentration in blood-time curve from 0 to τ at steady state
AUCtau,ss of D930(Sequence2) | 1day 0hour ~ 99day 0hour
  Area under the D930 concentration in blood-time curve from 0 to τ at steady
Cmax,ss of D565(Sequence1) | 1day 0hour ~ 99day 0hour
  The maximum D565 concentration between 0 and τ at steady state
Cmax,ss of D930(Sequence1) | 8day 0hour ~ 99day 0hour
  The maximum D930 concentration between 0 and τ at steady state
Cmax,ss of D565(Sequence2) | 96day 0hour ~ 99day 0hour
  The maximum D565 concentration between 0 and τ at steady state
Cmax,ss of D930(Sequence2) | 1day 0hour ~ 99day 0hour
  The maximum D930 concentration between 0 and τ at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine and Hospital, Seoul, South Korea